CLINICAL TRIAL: NCT03886493
Title: Neoadjuvant Dupilumab in Men With Localized High-Risk Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual due to COVID-19 pandemic.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J18116; IRB00182718 (Other: JHM IRB)
Record Dates: First submitted 2019-03-20; First posted 2019-03-22 (Actual); Results first posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-09

CONDITIONS: Prostate Cancer
Keywords: high-risk prostate cancer; localized prostate cancer; prior to prostatectomy; neoadjuvant
MeSH Terms: conditions — Prostatic Neoplasms | interventions — dupilumab

STUDY DESIGN:
Intervention Model Description: Men will be treated with dupilumab 600 mg s.q. on day 1, and then 300 mg s.q. on days 8,15, 22, 29, 36, 43. They will then undergo surgery on day 57. Fourteen days after the last dose of Dupixent, prostate glands will be harvested at the time of radical prostatectomy, and prostate tissue will be examined for the secondary endpoints. Follow-up evaluation for adverse events will occur 30 days and 60 days after surgery. Patients will then be followed by their urologists according to standard institutional practices, but will require PSA evaluations every 3 (±1) months during year 1 and every 6 (±2) months during years 2-3.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dupixent Subcutaneous (SQ) Injection (Experimental): Participants will be treated with dupilumab 600 mg SQ on day 1, and then 300 mg SQ on days 8,15, 22, 29, 36, 43. They will then undergo surgery on day 57. 14 days after the last dose of Dupixent, prostate glands will be harvested at the time of radical prostatectomy, and prostate tissue will be examined for the secondary endpoints.
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Dupilumab — dupilumab 600 mg SQ on day 1, and then 300 mg SQ on days 8,15, 22, 29, 36, 43.
  Other Names: Dupixent

SUMMARY:
This is a single-center, single arm, open-label phase II study evaluating the safety, anti-tumor effect, and immunogenicity of neoadjuvant Dupixent given prior to radical prostatectomy.

DETAILED DESCRIPTION:
This is a single-center, single arm, open-label phase II study evaluating the safety, anti-tumor effect, and immunogenicity of neoadjuvant Dupixent given prior to radical prostatectomy in men with high-risk localized prostate cancer (this trial will enroll men with at least high risk prostate cancer defined by NCCN Guidelines Version 2.2017 = clinical stage ≥T3a or PSA >20 ng/mL or Gleason score ≥8).

Patients will be recruited from the outpatient Urology clinic. Men will be treated with dupilumab 600 mg subcutaneously (SQ) on day 1, and then 300 mg SQ on days 8,15, 22, 29, 36, 43. They will then undergo surgery on day 57. 14 days after the last dose of Dupixent, prostate glands will be harvested at the time of radical prostatectomy, and prostate tissue will be examined for the secondary endpoints.

Follow-up evaluation for adverse events will occur 30 days and 60 days after surgery. Patients will then be followed by their urologists according to standard institutional practices, but will require PSA evaluations every 3 (±1) months during year 1 and every 6 (±2) months during years 2-3.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for this study, patients must meet all of the following criteria:

* Histologically confirmed adenocarcinoma of the prostate (clinical stage T1c-T3b, N0, M0) without involvement of lymph nodes, bone, or visceral organs
* Initial prostate biopsy is available for central pathologic review, and is confirmed to show at least 2 positive cores and a Gleason sum of ≥7
* Radical prostatectomy has been scheduled at Johns Hopkins Hospital
* Age ≥18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1, or Karnofsky score ≥ 70%
* Adequate bone marrow, hepatic, and renal function:

  * WBC >3,000 cells/mm3
  * ANC >1,500 cells/mm3
  * Hemoglobin >9.0 g/dL
  * Platelet count >100,000 cells/mm3
  * Serum creatinine <3 × upper limit of normal (ULN)
  * Serum bilirubin <3 × ULN
  * ALT <5 × ULN
  * AST <5 × ULN
  * Alkaline phosphatase <5 × ULN
* Willingness to provide written informed consent and HIPAA authorization for the release of personal health information, and the ability to comply with the study requirements (note: HIPAA authorization will be included in the informed consent)
* Willingness to use barrier contraception from the time of first dose of DUPILUMAB until the time of prostatectomy.

Exclusion Criteria:

To be eligible for this study, patients should not meet any of the following criteria:

* Presence of known lymph node involvement or distant metastases
* Other histologic types of prostate cancers such as ductal, sarcomatous, lymphoma, small cell, and neuroendocrine tumors
* Prior radiation therapy, hormonal therapy, biologic therapy, or chemotherapy for prostate cancer
* Prior immunotherapy/vaccine therapy for prostate cancer
* Concomitant treatment with other hormonal therapy or 5α-reductase inhibitors
* Current use of systemic corticosteroids or use of corticosteroids within 4 weeks of enrollment (inhaled corticosteroids for asthma or COPD are permitted)
* Use of experimental agents for prostate cancer within the past 3 months from time of screening
* History or presence of autoimmune disease requiring systemic immunosuppression (including but not limited to: inflammatory bowel disease, systemic lupus erythematosus, vasculitis, rheumatoid arthritis, scleroderma, multiple sclerosis, hemolytic anemia, Sjögren syndrome, and sarcoidosis)
* History of malignancy within the last 3 years, with the exception of non-melanoma skin cancers and superficial bladder cancer
* Uncontrolled major active infectious, cardiovascular, pulmonary, hematologic, or psychiatric illnesses that would make the patient a poor study candidate
* Known prior or current history of HIV and/or hepatitis B/C
* Significant eye disease

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Subjects must have a prostate in order to be eligible for this trial.
Enrollment: 7 (Actual)
Dates: Start 2019-08-28 (Actual); Primary Completion 2020-10-06 (Actual); Study Completion 2020-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Pienta, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dupixent Subcutaneous (SQ) Injection
Started | 7
Completed | 6
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Dupixent Subcutaneous (SQ) Injection
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in M2-TAM Infiltration From Baseline
Description: Change in M2-TAM infiltration (number of macrophages / cell nuclei per high power field [hpf]) measured in pre- dupilumab biopsy to M2-TAM infiltration measured in post-dupilumab specimen collected at time of radical prostatectomy (up to 59 days post-intervention). Degree of TAM infiltration will be analyzed using immunohistochemical staining for CD206. It is hypothesized that a positive value will be associated with better outcome and a negative value will reflect a worse outcome.
Time Frame: change from baseline to up to 59 days post-intervention
Population: Data could not be collected for this outcome measure due to COVID-19 pandemic restrictions.
Arm/Group | Dupixent Subcutaneous (SQ) Injection
Number analyzed (Participants) | 0

2. Secondary Outcome: Safety as Assessed by Number of Participants Experiencing Adverse Events
Description: Adverse events defined by NCI Common Toxicity Criteria version 4.0 (NCI CTCAE v4.0)
Time Frame: up to 59 days post-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Dupixent Subcutaneous (SQ) Injection
Number analyzed (Participants) | 7
Participants | 7

3. Secondary Outcome: Feasibility as Assessed by Number of Participants Who Have an Average Blood Loss in Excess of 2500 mL During Prostatectomy
Time Frame: up to 59 days post-intervention
Population: Only 6/7 participants had a prostatectomy.
Measure: Count of Participants; unit: Participants
Arm/Group | Dupixent Subcutaneous (SQ) Injection
Number analyzed (Participants) | 6
Participants | 0

4. Secondary Outcome: Feasibility as Assessed by Number of Participants With Average Prostatectomy Operative Time in Excess of 3.5 Hours
Time Frame: up to 59 days post-intervention
Population: Only 6/7 participants had a prostatectomy.
Measure: Count of Participants; unit: Participants
Arm/Group | Dupixent Subcutaneous (SQ) Injection
Number analyzed (Participants) | 6
Participants | 2

5. Secondary Outcome: Feasibility as Assessed by Number of Participants With Average Hospital Stay in Excess of 4 Days Post-prostatectomy
Time Frame: up to 59 days post-intervention
Population: Only 6/7 participants had a prostatectomy
Measure: Count of Participants; unit: Participants
Arm/Group | Dupixent Subcutaneous (SQ) Injection
Number analyzed (Participants) | 6
Participants | 0

6. Secondary Outcome: CD8+ T-cell Infiltration in Post-treatment Prostate Glands
Description: mean CD4+ T-cell staining percentage and CD4+/Treg ratio in harvested tumor tissue collected from prostatectomy specimen
Time Frame: up to 59 days post-intervention
Population: Data could not be collected for this outcome measure due to COVID-19 pandemic restrictions.
Arm/Group | Dupixent Subcutaneous (SQ) Injection
Number analyzed (Participants) | 0

7. Secondary Outcome: CD4+ T-cell and Treg Infiltration in Post-treatment Prostate Glands
Description: as for outcome 6
Time Frame: up to 59 days post-intervention
Population: Data could not be collected for this outcome measure due to COVID-19 pandemic restrictions.
Arm/Group | Dupixent Subcutaneous (SQ) Injection
Number analyzed (Participants) | 0

8. Secondary Outcome: Expression of Apoptosis Marker (Annexin V) in Post-treatment Prostate Tumor Specimen as Measured by Mean Staining Percentage in Tumor Tissue
Description: Mean staining percentage of Annexin V in tumor tissue, using TUNEL (Terminal deoxynucleotidyl transferase dUTP nick end labeling) staining.
Time Frame: up to 59 days post-intervention
Population: Data could not be collected for this outcome measure due to COVID-19 pandemic restrictions.
Arm/Group | Dupixent Subcutaneous (SQ) Injection
Number analyzed (Participants) | 0

9. Secondary Outcome: Expression of Cell Proliferation in Post-treatment Prostate Tumor Specimen as Measured by Mean Staining Percentage of Ki-67 in Tumor Tissue
Time Frame: up to 59 days post-intervention
Population: Data could not be collected for this outcome measure due to COVID-19 pandemic restrictions.
Arm/Group | Dupixent Subcutaneous (SQ) Injection
Number analyzed (Participants) | 0

10. Secondary Outcome: Proportion of Participants With Pathological Complete Response
Description: Pathological response is defined as the absence of tumor identification by study pathologist on standard histological analysis of resected prostate specimens.
Time Frame: 1 month post-prostatectomy
Population: Data could not be collected for this outcome measure due to COVID-19 pandemic restrictions.
Arm/Group | Dupixent Subcutaneous (SQ) Injection
Number analyzed (Participants) | 0

11. Secondary Outcome: Proportion of Participants Who Achieve an Undetectable PSA at 2 Months Post-prostatectomy
Description: Proportion of participants with PSA <0.1ng/mL by 2 months after prostatectomy
Time Frame: 2 months post-prostatectomy
Population: Data could not be collected for this outcome measure due to COVID-19 pandemic restrictions.
Arm/Group | Dupixent Subcutaneous (SQ) Injection
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: up to 1 year
Arm/Group | Dupixent Subcutaneous (SQ) Injection
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 7/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dupixent Subcutaneous (SQ) Injection (N=7)
Urinary incontinence (Renal and urinary disorders) | 5 (5)
Headache, intermittent (General disorders) | 2 (2)
Bloating (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
edema in right calf and ankle (Blood and lymphatic system disorders) | 1 (1)
elevated hemoglobin (Blood and lymphatic system disorders) | 1 (1)
eye pain (Eye disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Vivid dreams (General disorders) | 1 (1)
hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Increased creatinine (Renal and urinary disorders) | 1 (1)
induration at injection site on abdomen (Skin and subcutaneous tissue disorders) | 1 (1)
laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
loss of appetite (Metabolism and nutrition disorders) | 1 (1)
maculo papular rash on abdomen (Skin and subcutaneous tissue disorders) | 2 (2)
nausea (Gastrointestinal disorders) | 1 (1)
pruritis at site of injection on abdomen (Skin and subcutaneous tissue disorders) | 1 (1)
reproductive system disorder, other blood in ejaculate (Reproductive system and breast disorders) | 1 (1)
Right AC bruising related to blood draw (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration upper lip (Skin and subcutaneous tissue disorders) | 1 (1)
toothache (Gastrointestinal disorders) | 1 (1)
urinary retention (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-03): https://cdn.clinicaltrials.gov/large-docs/93/NCT03886493/Prot_SAP_000.pdf